CLINICAL TRIAL: NCT04369053
Title: Prevention of Colorectal Cancer Through Multiomics Blood Testing
Acronym: PREEMPT CRC
Status: Completed | Type: Observational
Sponsor: Freenome Holdings Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FRNM-004
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Colon Cancer; Rectal Cancer; Colon Neoplasm; Colon Diseases; Colon Lesion; Colon Polyp; Colorectal Cancer; Polyp; Adenoma; Rectal Diseases; Gastrointestinal Tract Cancers
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colonic Diseases; Colonic Polyps; Colorectal Neoplasms; Polyps; Adenoma; Rectal Diseases; Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens will be de-identified and used to validate the performance characteristics of the Freenome test.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Freenome test — Participants who provide informed consent, meet the eligibility criteria and provide a blood sample for this study will be enrolled. Participants will undergo blood collection and will then complete a standard-of-care screening colonoscopy.
  Other Names: Single Group Assignment

SUMMARY:
The PREEMPT CRC study is a prospective multi-center observational study to validate a blood-based test for the early detection of colorectal cancer by collecting blood samples from average-risk participants who will undergo a routine screening colonoscopy.

DETAILED DESCRIPTION:
Freenome is using a type of artificial intelligence, called machine learning, to identify patterns of cell-free biomarkers in blood to detect cancer early. The purpose of this prospective multi-center observational study is to validate a blood-based test for the detection of colorectal cancer by collecting blood samples from average-risk participants who will undergo a routine screening colonoscopy.

ELIGIBILITY:
Key Inclusion Criteria

1. 45-85 years of age
2. Willing to undergo a standard-of-care screening colonoscopy
3. Able and willing to provide a blood sample
4. Able and willing to sign informed consent

Key Exclusion Criteria

1. Known hereditary gastrointestinal cancer syndrome (for example, hereditary non-polyposis CRC syndrome (HNPCC) or Lynch syndrome, or familial adenomatous polyposis (FAP)
2. Personal history 2.1 CRC or colorectal adenoma 2.2 Inflammatory bowel disease (IBD), including chronic ulcerative colitis (CUC) and crohn's disease (CD) 2.3 Colonoscopy in the 9 years preceding enrollment 2.4 Stool DNA testing in the 2 years preceding enrollment 2.5 Symptoms of lower gastrointestinal tract disease warranting colonoscopic evaluation
3. A medical condition which, in the opinion of the Investigator, should preclude enrollment in the study
4. Participated or currently participating in a clinical research study in which an experimental medication has been administered during the 60 days up to and including the date of providing informed consent or may be administered through the time of the colonoscopy

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants aged between 45 and 85 who are eligible for CRC screening and scheduled for a standard-of-care screening colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 48995 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aasma Shaukat, MD, MPH, Principal Investigator — NYU Langone Health; Theodore R Levin, MD, Principal Investigator — Kaiser Permanente Division of Research
Locations (148):
- United States (147):
  - Central Alabama Research, Birmingham, Alabama
  - Alabama Oncology, Birmingham, Alabama
  - Clinical Research Associates, Huntsville, Alabama
  - Del Sol Research Management, Chandler, Arizona
  - Honor Health, Scottsdale, Arizona
  - Del Sol Research Management,, Tucson, Arizona
  - Preferred Research Partners, Little Rock, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Precision Research Institute, Chula Vista, California
  - John Muir Health, Concord, California
  - Carbon Health, Corona, California
  - Miller Bioconnect, El Cajon, California
  - Gastroenterology and Liver Institute, Escondido, California
  - Women's Cancer Network, Fresno, California
  - San Diego Clinical Trials, La Mesa, California
  - Urology Alliance Clinical Research, Los Angeles, California
  - Science 37, Los Angeles, California
  - Mercy Cancer Center, Merced, California
  - Diverse Research Solutions, Oxnard, California
  - Pomona Valley Hospital Medical Center/Cancer Care Center, Pomona, California
  - St. Mary's Medical Center, San Francisco, California
  - Dominican Hospital Dignity Health, Santa Cruz, California
  - Stockton Hematology Oncology, Stockton, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Gastroenterology Associates of Fairfield County, Bridgeport, Connecticut
  - Eastern CT Hematology and Oncology Associates, Norwich, Connecticut
  - Stamford Hospital, Stamford, Connecticut
  - RecioMed Clinical Research, Boynton Beach, Florida
  - Hillcrest Medical Research, DeLand, Florida
  - Universal Axon Clinical Research, Doral, Florida
  - Palmetto Research, Hialeah, Florida
  - Clinical Research of Homestead, Homestead, Florida
  - I.H.S Health, LLC, Kissimmee, Florida
  - Mid Florida Hematology & Oncology Center, Orange City, Florida
  - Advanced Gastroenterology Associates, LLC, Palm Harbor, Florida
  - Emerald Coast OBGYN, Panama City, Florida
  - Ascension Sacred Heart, Pensacola, Florida
  - United Medical Research, Port Orange, Florida
  - Charter Research, The Villages, Florida
  - Morehouse School of Medicine, Atlanta, Georgia
  - Crisp Regional Hospital, Cordele, Georgia
  - Cancer Center of Middle Georgia (QCCA), Dublin, Georgia
  - SpeciCare, Inc, Gainesville, Georgia
  - Specicare, Gainesville, Georgia
  - University of Chicago, Chicago, Illinois
  - Walgreens, Deerfield, Illinois
  - Silver Cross Hospital and Medical centers, Orland Park, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Rockford Gastroenterology, Rockford, Illinois
  - Northwest Oncology & Hematology, Rolling Meadows, Illinois
  - Springfield Clinic, LLP, Springfield, Illinois
  - Margaret Mary, Batesville, Indiana
  - Objective Health Network (Digestive Research Alliance of Michiana, LLC), South Bend, Indiana
  - Aton Health, Leawood, Kansas
  - Ascension Via Christi Hospital, Wichita, Wichita, Kansas
  - Ascension Via Christi Wichita, Wichita, Kansas
  - Saint Joseph Cancer Center, Lexington, Kentucky
  - Delta Research Partners, Bastrop, Louisiana
  - New Orleans Research Institute, Metairie, Louisiana
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Louisiana Research Center, Shreveport, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Ascension St. Agnes Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Commonwealth Clinical Studies, Brockton, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health, Detroit, Michigan
  - Ascension Providence Rochester Hospital, Rochester Hills, Michigan
  - Covenant HealthCare, Saginaw, Michigan
  - Allina Health Cancer Institute, Minneapolis, Minnesota
  - University of Minnesota, School of Public Health, Environmental Health Sciences, Minneapolis, Minnesota
  - Winona Health System, Winona, Minnesota
  - Memorial Hospital at Gulfport, Gulfport, Mississippi
  - Central Care Cancer Center, Bolivar, Missouri
  - Carroll County Memorial Hospital, Carrollton, Missouri
  - Hannibal Regional Hospital, Hannibal, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, North Kansas City, Missouri
  - Billings Clinic, Billings, Montana
  - Logan Health Research, Kalispell, Montana
  - Quality Clinical Research, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Cancer Care Specialists Reno, Reno, Nevada
  - Inspira Medical Center, Mullica Hill, New Jersey
  - St Joseph University, Paterson, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Our Lady of Lourdes Hospital, Binghamton, New York
  - NYU, New York, New York
  - NY Cancer & Blood Specialists, Port Jefferson Station, New York
  - White Plains Hospital, White Plains, New York
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cumberland Research Associates, Fayetteville, North Carolina
  - Wakemed, Raleigh, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Trial Management Associates, Wilmington, North Carolina
  - Altru Health System, Grand Forks, North Dakota
  - Gabrail Cancer Center Research, Canton, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Objective Health Network, Dayton, Ohio
  - Hightower Clinical Research, Oklahoma City, Oklahoma
  - Hightower Clinical, Oklahoma City, Oklahoma
  - St. Charles Health System, Inc, Bend, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Bloomsburg Hospital, Bloomsburg, Pennsylvania
  - Doylestown Health, Doylestown, Pennsylvania
  - Clinical Research Associates of Central PA, DuBois, Pennsylvania
  - Pennsylvania Cancer Specialists & Research Institute, Gettysburg, Pennsylvania
  - US Digestive Health at Lancaster, Lancaster, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Donald Guthrie Foundation, Sayre, Pennsylvania
  - Guthrie Medical Group, Sayre, Pennsylvania
  - USDH Clinical Research, Wyomissing, Pennsylvania
  - US Digestive Health at Wyomissing, Wyomissing, Pennsylvania
  - Cancer Care Associates of York (QCCA), York, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - MUSC, Charleston, South Carolina
  - MacLeod Center for Cancer Treatment and Research, Florence, South Carolina
  - McLeod Health, Florence, South Carolina
  - Carolina Blood and Cancer Care Associates, Rock Hill, South Carolina
  - Circle Clinical Research, Pierre, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - ObjectiveHealth, Inc, Franklin, Tennessee
  - The Jackson Clinic, PA, Jackson, Tennessee
  - The Jackson Clinic, Jackson, Tennessee
  - Elligo Health Research, Inc., Austin, Texas
  - Christus Spohn Shoreline Hospital, Corpus Christi, Texas
  - Horizon Clinical Research Group, Houston, Texas
  - Oncology Consultants, Houston, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Christus Trinity Mother Frances Health System, Tyler, Texas
  - Advanced Research Institute, Ogden, Utah
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - INOVA, Fairfax, Virginia
  - Verity Research Inc, Fairfax, Virginia
  - Centra Lynchburg Hematology Oncology, Lynchburg, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Washington Gastroenterology, Bellevue, Washington
  - Northwest Medical Specialties (QCCA), Tacoma, Washington
  - SSM Health-Dean Medical Group, Madison, Wisconsin
  - Ascension Columbia St. Mary's Wisconsin, Milwaukee, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Forzani and MacPhail Colon Cancer Screening Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shaukat A, Burke CA, Chan AT, Grady WM, Gupta S, Katona BW, Ladabaum U, Liang PS, Liu JJ, Putcha G, Robertson DJ, Schoen RE, Meng Z, Piscitello A, Sun CK, Xu C, Lin CJ, Lee LC, Baldo L, Levin TR; PREEMPT CRC Investigators. Clinical Validation of a Circulating Tumor DNA-Based Blood Test to Screen for Colorectal Cancer. JAMA. 2025 Jul 1;334(1):56-63. doi: 10.1001/jama.2025.7515. PMID 40455622
- [Derived] Kortlever TL, Ferlizza E, Lauriola M, Borrelli F, Porro A, Spaander MCW, Bossuyt PM, Ricciardiello L, Dekker E. Diagnostic Accuracy of an Add-On, Blood-Based Screening Test for Colorectal Cancer in Two Established Screening Programmes. Aliment Pharmacol Ther. 2025 Jun;61(12):1935-1943. doi: 10.1111/apt.70141. Epub 2025 Apr 10. PMID 40207404
- [Derived] Mills K, Figueroa F, Knight R, Ekpo E, Lee LC, Baldo L, Xu C, Wang S, Adelman RM, Pemu P, Levin T, Shaukat A, Liu JJ. Fact or Myth? Black Patients Do Not Want to Participate in Clinical Trials. Clin Transl Gastroenterol. 2025 Apr 1;16(4):e00826. doi: 10.14309/ctg.0000000000000826. PMID 39878425

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who met the eligibility criteria and signed the informed consent were enrolled in the study.
Pre-assignment Details: Of 48,995 subjects enrolled in the PREEMPT CRC study, 32,731 consecutively enrolled on or after a pre-specified cut-off date were included in the clinical validation cohort. 27,010 subjects from the clinical validation cohort were evaluable with confirmed clinical findings and valid blood test results.
Groups:
- Enrolled Subjects: Study subjects who were aged 45 to 85 years, asymptomatic, at average risk of colorectal cancer, and willing to undergo a standard-of-care screening colonoscopy.
Period: Overall Study
Arm/Group | Enrolled Subjects
Started | 48995
Completed | 27010
Not Completed | 21985
Not completed — Enrolled prior to the Pre-specified Cut-off Date | 16264
Not completed — Withdrawal by Subject | 773
Not completed — Lost to Follow-up | 182
Not completed — Blood Test and/or Colonoscopy Reasons | 4766

BASELINE CHARACTERISTICS:
Population: Subjects enrolled on or after the pre-specified cut-off date who had confirmed clinical findings and valid blood test results.
Groups:
- Evaluable Subjects: Subjects enrolled on or after the pre-specified cut-off date who had confirmed clinical findings and valid blood test results.
Arm/Group | Evaluable Subjects
Number analyzed (Participants) | 27010
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.1 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15076
  Male | 11934
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 78
  Asian | 2381
  Native Hawaiian or Other Pacific Islander | 72
  Black or African American | 3038
  White | 19707
  More than one race | 136
  Unknown or Not Reported | 1598
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3189
  Not Hispanic or Latino | 22421
  Unknown or Not Reported | 1400

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity for Colorectal Cancer
Description: Proportion of participants with a positive test result among those who had a diagnosis of colorectal cancer
Time Frame: 90 days
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Evaluable Subjects
Number analyzed (Participants) | 27010
Percent | 79.2 [68.4 to 86.9]

2. Primary Outcome: Specificity for Advanced Colorectal Neoplasia
Description: Proportion of participants with a negative test result among those who had non-advanced precancerous lesions or negative findings (non-neoplastic or no findings)
Time Frame: 90 days
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Evaluable Subjects
Number analyzed (Participants) | 27010
Percent | 91.5 [91.2 to 91.9]

3. Primary Outcome: Negative Predictive Value for Advanced Colorectal Neoplasia
Description: Proportion of participants with a diagnosis of non-advanced precancerous lesions or negative findings (non-neoplastic or no findings) among those who had a negative test result
Time Frame: 90 days
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Evaluable Subjects
Number analyzed (Participants) | 27010
Percent | 90.8 [90.7 to 90.9]

4. Primary Outcome: Positive Predictive Value for Advanced Colorectal Neoplasia
Description: Proportion of participants with a diagnosis of colorectal cancer or advanced precancerous lesions among those who had a positive test result
Time Frame: 90 days
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Evaluable Subjects
Number analyzed (Participants) | 27010
Percent | 15.5 [14.2 to 16.8]

5. Secondary Outcome: Sensitivity for Advanced Precancerous Lesion
Description: Proportion of participants with a positive test result among those who had a diagnosis of advanced precancerous lesions
Time Frame: 90 days
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Evaluable Subjects
Number analyzed (Participants) | 27010
Percent | 12.5 [11.3 to 13.8]

6. Other Pre Specified Outcome: Census-adjusted Sensitivity for Colorectal Cancer
Description: U.S. census sex- and age-adjusted sensitivity for colorectal cancer Proportion of participants with a positive test result among those who had a diagnosis of colorectal cancer
Time Frame: 90 days
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Evaluable Subjects
Number analyzed (Participants) | 27010
Percent | 81.1 [71.3 to 88.1]

7. Other Pre Specified Outcome: Census-adjusted Specificity for Advanced Colorectal Neoplasia
Description: U.S. census sex- and age-adjusted specificity for advanced colorectal neoplasia Proportion of participants with a negative test result among those who had non-advanced precancerous lesions or negative findings (non-neoplastic or no findings)
Time Frame: 90 days
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Evaluable Subjects
Number analyzed (Participants) | 27010
Percent | 90.4 [90.0 to 90.7]

8. Other Pre Specified Outcome: Census-adjusted Negative Predictive Value for Advanced Colorectal Neoplasia
Description: U.S. census sex- and age-adjusted negative predictive value for advanced colorectal neoplasia Proportion of participants with a diagnosis of non-advanced precancerous lesions or negative findings (non-neoplastic or no findings) among those who had a negative test result
Time Frame: 90 days
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Evaluable Subjects
Number analyzed (Participants) | 27010
Percent | 90.5 [90.4 to 90.7]

9. Other Pre Specified Outcome: Census-adjusted Positive Predictive Value for Advanced Colorectal Neoplasia
Description: U.S. census sex- and age-adjusted positive predictive value for advanced colorectal neoplasia Proportion of participants with a diagnosis of colorectal cancer or advanced precancerous lesions among those who had a positive test result
Time Frame: 90 days
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Evaluable Subjects
Number analyzed (Participants) | 27010
Percent | 15.5 [14.3 to 16.7]

10. Other Pre Specified Outcome: Census-adjusted Sensitivity for Advanced Precancerous Lesion
Description: U.S. census sex- and age-adjusted sensitivity for advanced precancerous lesion Proportion of participants with a positive test result among those who had a diagnosis of advanced precancerous lesions
Time Frame: 90 days
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Evaluable Subjects
Number analyzed (Participants) | 27010
Percent | 13.7 [12.4 to 15.0]

ADVERSE EVENTS:
Time Frame: Twenty-four hours within the study blood collection
Description: Pre-specified to only collect adverse events related to study blood collection
Groups:
- Safety Analysis Set: Subjects with attempted blood collection
Arm/Group | Safety Analysis Set
All-Cause Mortality (participants affected / at risk) | 0/31888
Serious Adverse Events (participants affected / at risk) | 0/31888
Other Adverse Events (participants affected / at risk) | 83/31888
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Analysis Set (N=31888)
Dizziness, syncope, contusion, and other observed minor complications (General disorders) | 83

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At Sponsor's request, the PI shall remove any Confidential Information (other than Study Results) prior to submitting or presenting the materials. Upon Sponsor's request, PI shall further delay publication or presentation for x period of days to allow Sponsor to protect its interests in any Sponsor Inventions described in any materials.

DOCUMENTS (2):
  • Study Protocol (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT04369053/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT04369053/SAP_001.pdf